CLINICAL TRIAL: NCT00398593
Title: Patient Adherence to Prescribed Therapy in Ulcerative Colitis: an Investigation of Barriers & Methods of Improvement.
Brief Title: Methods of Improvement Adherence With Therapy in Ulcerative Colitis.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Carolyn Burden, Leicester General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UHL 09788; REC 06/Q2502/100
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Ulcerative Colitis
Keywords: Adherence with therapy; Adherence enhancing intervention; Nonadherence; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Adherence Interventions

INTERVENTIONS:
Behavioral: Range of electronic pill dispensers with alarms — Patients will be offered 1. Counselling with education and/or 2. Electronic reminders

SUMMARY:
Ulcerative Colitis is associated with a significantly increased risk of colorectal cancer. This risk can be reduced through regular medication with 5ASA compounds. Their effectiveness however is limited by poor adherence to the treatment protocols by many patients.

The hypothesis which underlies this proposal is that if the factors responsible for poor compliance can be identified, interventions could be developed which would help to overcome the barriers which exist in individual patients. These interventions would be based on the reasons for non-adherence, specifically tailored to the needs of the individual. As a result such interventions will improve patients' adherence with prescribed 5ASA and therefore reduce the relapses of the disease and a cancer risk.

DETAILED DESCRIPTION:
Poor adherence to treatment is well recognised and significantly contributes to treatment failures. In ulcerative colitis it may be associated with an increased risk of colorectal cancer. Estimates for non-adherence range from 15% to 93% with an average of around a third of patients failing to adhere to their recommended therapeutic regimen.

The study aims to evaluate a wide-ranging approach to reducing poor adherence, which is based on factors associated with non-adherence and involves the patient in choosing interventions.

The effectiveness of the overall intervention will be assessed through a randomised controlled trial comparing intervention against standard care.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-80.
* Those in whom a diagnosis of ulcerative colitis is based on histological confirmation of the disease.
* Patients who are on daily maintenance therapy with 5 ASA medication.
* Patients who have read the information leaflet and voluntarily given informed consent.

Exclusion Criteria:

* Those aged under 18 years old.
* Those with a diagnosis of Crohn's disease.
* Patients not on regular 5ASA compound as maintenance therapy.
* Patients unable to give informed consent.
* Patients who do not wish to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Levels of patient adherence to therapy will be assessed in two ways: | 1 year
through pill counts and measurement of salicylate levels in urine samples. | 1 year

SECONDARY OUTCOMES:
Quantitative data will be collected through feedback from patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John F Mayberry, DScMD, Principal Investigator — University Hospitals, Leicester

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391